CLINICAL TRIAL: NCT06360328
Title: Success Rates of Video- vs. Direct Laryngoscopy for Endotracheal Intubation in Anesthesiology Residents: A Randomized Controlled Trial" (The JuniorDoc-VL-Trial)
Acronym: JuniorDoc-VL
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital Heidelberg (Other)
Responsible Party: Principal Investigator, Dr. med. Davut Deniz Uzun, Medical Doctor, Post-Doc Researcher, Department of Anesthesiology, University Hospital Heidelberg
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 033-2024
Record Dates: First submitted 2024-04-08; First posted 2024-04-11 (Actual); Last update posted 2025-01-22 (Actual); Status verified 2025-01

CONDITIONS: Intubation Complication; Intubation
Keywords: Airway Management; Video-Laryngoscopy; First-Pass-Success; Skill of Intubation; Direct Laryngoscopy

STUDY DESIGN:
Intervention Model Description: Control group = direct laryngoscopy Intervention group = video laryngoscopy
Who Masked: Participant
Masking Description: Only the patient is blinded, as the participants (residents) cannot be blinded.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- direct Laryngoscopy (No Intervention): The resident intubates using direct laryngoscopy .
- video Laryngoscopy (Experimental): The resident intubates using video laryngoscopy
  Interventions: Device: video laryngoscopy

INTERVENTIONS:
Device: video laryngoscopy — The residents used video laryngoscopy for endotracheal intubation
  Arms: video Laryngoscopy

SUMMARY:
Securing the airway through endotracheal intubation (ETI) is a fundamental skill for anaesthetists. It is used during surgery, in the intensive care unit, during periprocedural anaesthesia and in emergency medicine. The clinical relevance of airway management is demonstrated in particular by the fact that the main cause of serious anaesthesia-related complications lies in the area of airway management. increasing technological developments in recent years (e.g. video laryngoscopy [VL]) aim to reduce the complication rate in the area of airway management. however, there are currently a large number of VLs available, which differ massively in their application. Therefore, it is essential to systematically collect data and develop structured training in airway management, taking into account current technological developments.While endotracheal intubation is traditionally performed with a direct laryngoscope, indirect video laryngoscopy, with chip-based camera technology at its tip, has been introduced across the board in recent years and is now part of standard clinical and preclinical equipment. Doctors in advanced training are trained with a focus on direct laryngoscopy; the use of and training in indirect video laryngoscopy does not follow any standards; in addition, the decision as to which method of securing the airway is chosen has so far been the responsibility of the individual doctor in anaesthesiology, although there is a tendency for the VL to be associated with a higher success rate in the first intubation attempt, the so-called "first-pass success".The main aim of this clinical prospective, randomised controlled trial is to train anaesthetists in advanced training in conventional direct laryngoscopy on the one hand and indirect video laryngoscopy (VL) on the other, with a focus on tracking the progress of their skills after 200 intubations with regard to first-pass success.

DETAILED DESCRIPTION:
Securing the airway is a core competence of anaesthetists, intensive care physicians and emergency physicians, as oxygenation of the human organism is not possible without an open or secured airway. The introduction of new techniques and the implementation of guidelines and strategies for the care of the difficult airway have contributed significantly to a reduction in morbidity and mortality. Of particular importance are problems that can occur during airway management, which are referred to in anaesthesiology as the "difficult airway". The term "difficult airway" refers to problems that can occur during airway management. Despite technological advances in the field of airway management, such as the use of video laryngoscopes, the definition of a difficult airway is still based on the traditional methods of mask ventilation and intubation using direct laryngoscopy. In recent years, several airway management studies suggest that the primary use of video laryngoscopes in adult patients undergoing endotracheal intubation is associated with a reduction in failed attempts and complications such as hypoxaemia.Problems during endotracheal intubation are often subsumed under the term "difficult intubation" without differentiating between "laryngoscopy" and "endotracheal intubation". However, if indirect laryngoscopy techniques are used, such as videolaryngoscopic intubation, a clear distinction must be made between the two procedures, as the incidence of difficult laryngoscopy is always lower than that of difficult or impossible intubation. The incidence of difficult direct laryngoscopy is 1.5% to 8.0%, while the incidence of difficult intubation is slightly lower. A potentially life threatening unexpected "cannot intubate, cannot ventilate" situation has a probability of0.008% (1:13,000) to 0.004% (1:25,000). In a randomised study design, we would like to record resident anaesthesiologists (first-year) learning the skill of endotracheal intubation with direct and indirect laryngoscopy in order to derive and analyse anaesthesiological quality parameters, such as first-pass success and possible complications. The individual learning curves of those entering the profession will also be taken into account in order to gain insights for the improvement of training programmes and training methods in anaesthesiology.

ELIGIBILITY:
Inclusion Criteria:

* First Year Anesthesiology Residents

Exclusion Criteria:

* Physicians' refusal to participate in the study
* Participants in another study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2024-04-01 (Actual); Primary Completion 2027-04-01 (Estimated); Study Completion 2027-08-01 (Estimated)

PRIMARY OUTCOMES:
Rate of Successful tracheal intubation on the first attempt (First-Pass-Success). | Directly during intubation
  Rate of Successful tracheal intubation on the first attempt (First-Pass-Success).

SECONDARY OUTCOMES:
Number of complications such as desaturation below 90% Oxygen saturation level (SpO2), regurgitation, dental or soft tissue trauma. | Directly during intubation
  Number of complications such as desaturation below 90% Oxygen saturation level (SpO2), regurgitation, dental or soft tissue trauma.
Specify the number of attempts made during laryngoscopy. | Directly during intubation
  Specify the number of attempts made during laryngoscopy.
Compare the level of training with intubation success. | During the analysis
  Compare the level of training with intubation success.
Mention any failures or transitions to other rescue techniques. | Directly during intubation
  Mention any failures or transitions to other rescue techniques.
Specify the use of Optimal External Laryngeal Manipulation (OELM) techniques such as backward, upward and rightward pressure (BURP) Cricoid Pressure (CP) or adjustment of the participant's head and neck position. | Directly during intubation
  Specify the use of Optimal External Laryngeal Manipulation (OELM) techniques such as backward, upward and rightward pressure (BURP) Cricoid Pressure (CP) or adjustment of the participant's head and neck position.
When using VL, record the occurrence of fogging. | Directly during intubation
  When using VL, record the occurrence of fogging.
Assess the glottic view using the Cormack-Lehane-Score (I - IV). (I = good view) | Directly during intubation
  Assess the glottic view using the Cormack-Lehane-Score (I - IV).(I = good view)
assess the glottic view using the Percentage of Glottic Opening Score (POGO) (0%-100%). (0%= no view, 100% best view) | Directly during intubation
  assess the glottic view using the Percentage of Glottic Opening Score (POGO) (0%-100%)(0%= no view, 100% best view)

CONTACTS AND LOCATIONS:
Overall Officials: Davut Deniz Uzun, Dr. / MD, Principal Investigator — University of Heidelberg, Medical Faculty, Departement of Anesthesiology, Heidelberg, Germany
Locations (1):
- Medical Faculty Heidelberg, Department of Anesthesiology, Heidelberg University,, Heidelberg, Baden-Wurttemberg, Germany

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Uzun DD, Eicher S, Mohr S, Weigand MA, Schmitt FCF. Success rates of video vs. direct laryngoscopy for endotracheal intubation in anesthesiology residents: a study protocol for a randomized controlled trial (JuniorDoc-VL-Trial). Trials. 2025 Feb 27;26(1):75. doi: 10.1186/s13063-025-08785-y. PMID 40016759